CLINICAL TRIAL: NCT04904913
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of IBI362 in Chinese Overweight and Obese Subjects
Brief Title: A Study of IBI362 Evaluating Weight Loss in Obese and Overweight Chinese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI362B201
Record Dates: First submitted 2021-05-25; First posted 2021-05-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Overweight/ Obesity
MeSH Terms: interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- IBI362 high dose (Experimental): high dose IBI362 administered subcutaneously (SC) once a week.
  Interventions: Drug: IBI362
- IBI362 low dose (Experimental): Low dose IBI362 administered subcutaneously (SC) once a week.
  Interventions: Drug: IBI362
- placebo (Placebo Comparator): placebo administered subcutaneously (SC) once a week.
  Interventions: Other: placebo
- IBI362 moderate dose (Experimental): moderate dose IBI362 administered subcutaneously (SC) once a week.
  Interventions: Drug: IBI362
- IBI362 extra high dose (Experimental): extra high dose IBI362 administered subcutaneously (SC) once a week.
  Interventions: Drug: IBI362

INTERVENTIONS:
Drug: IBI362 — IBI362 administered subcutaneously (SC) once a week.
  Arms: IBI362 extra high dose; IBI362 high dose; IBI362 low dose; IBI362 moderate dose
Other: placebo — placebo administered subcutaneously (SC) once a week.
  Arms: placebo

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled study conducted in overweight or obese subjects. This study is divided into the first stage and the second stage. The participant enrollment and data analysis in the two stage are independent and do not influence each other.

In the first stage of this study, about 240 subjects will be enrolled. Qualified subjects will receive placebo in a 2-week introduction period, after that, they will be randomized to IBI362 low dose, IBI362 moderate dose, IBI362 high dose groups, in every group, subjects will be randomized to IBI362 and placebo groups at a ratio of 3:1. Random stratification is performed based on BMI < 28.0 kg/㎡ and BMI≥28.0 kg/㎡. The subjects received drug administration once weekly. The entire trial covers a 3-week screening period, a 2-week placebo introduction period, a-24 week double-blind treatment period, and a 12-week drug discontinuation follow-up period. During the entire research period, the subjects shall maintain diet and exercise control.

The second stage is IBI362 extra high dose study, about 80 subjects will be enrolled. Qualified participants will receive placebo in a 2-week introduction period, after that, they will be randomized to IBI362 extra high dose and placebo groups at a ratio of 3:1. The subjects received drug administration once weekly. The entire trial covers a 3-week screening period, a 2-week placebo introduction period, a 24-week double-blind treatment period, a 24-week extended treatment period, and a 12-week drug discontinuation follow-up period. The 24-week extended treatment period is optional. During the entire research period, the subjects shall maintain diet and exercise control.

ELIGIBILITY:
Inclusion Criteria:

1. The first stage: Body mass Index (BMI) ≥28 kilograms per square meter (kg/m²), or ≥24 kg/m² with at least one of the following comorbidities: hyperphagia, pre-diabetes, hypertension, dyslipidemia, fatty liver disease, weight-bearing joint pain, obesity-induced dyspnea or obstructive sleep apnea syndrome; The second stage: Body mass Index (BMI) ≥30 kilograms per square meter (kg/m²)
2. The weight change of the subjects before and after the introduction period was less than 5.0%

Exclusion Criteria:

1. Diabetes mellitus
2. Weight change > 5.0% after diet and exercise control for at least 12 weeks before screening
3. Have used or are currently using weight loss drugs within 3 months before screening
4. History of pancreatitis
5. Family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
6. History of moderate to severe depression，or have a history of serious mental illness
7. Any lifetime history of a suicide attempt

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline ,week 24
  Percent Change from Baseline in Body Weight

SECONDARY OUTCOMES:
Percentage of Participants who Achieve ≥5% Body Weight Reduction | Baseline, Week 24
Percentage of Participants who Achieve ≥10% Body Weight Reduction | Baseline, Week 24
Absolute change from Baseline in body weight | Baseline, Week 24
Change from Baseline in Waist Circumference | Baseline, Week 24
Change from Baseline in BMI | Baseline, Week 24
Change from Baseline in HbA1c | Baseline, Week 24
Change from Baseline in fasting plasma glucose | Baseline, Week 24
Change from Baseline in systolic blood pressure | Baseline, Week 24
Change from Baseline in diastolic blood pressure | Baseline, Week 24
Change from Baseline in total cholesterol | Baseline, Week 24
Change from Baseline in low-density lipoprotein cholesterol | Baseline, Week 24
Change from Baseline in high-density lipoprotein cholesterol | Baseline, Week 24
Change from Baseline in triglyceride | Baseline, Week 24
Change from Baseline in serum uric acid | Baseline, Week 12, Week 24
Change from Baseline in IWQoL-Lite-CT questionnaire scores | Baseline, Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University people's hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ji L, Jiang H, Cheng Z, Qiu W, Liao L, Zhang Y, Li X, Pang S, Zhang L, Chen L, Yang T, Li Y, Qu S, Wen J, Gu J, Deng H, Wang Y, Li L, Han-Zhang H, Ma Q, Qian L. A phase 2 randomised controlled trial of mazdutide in Chinese overweight adults or adults with obesity. Nat Commun. 2023 Dec 14;14(1):8289. doi: 10.1038/s41467-023-44067-4. PMID 38092790